CLINICAL TRIAL: NCT06826040
Title: A Phase 1 Clinical Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-tumor Activity of SKB445 for Injection in Patients With Advanced Solid Tumors
Brief Title: SKB445 for Injection in Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB445-I-01
Record Dates: First submitted 2025-01-19; First posted 2025-02-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation Phase (Experimental): Subject will be dosed with SKB445 for injection q3w
  Interventions: Drug: SKB445 for injection

INTERVENTIONS:
Drug: SKB445 for injection — SKB445 for injection is administered every 3 weeks (q3w) until radiographic disease progression (PD), intolerable toxicity, death, or discontinuation of treatment, whichever occurs first.

SUMMARY:
This is a multicenter, open-label, multiple-dose dose finding and expansion study to evaluate the safety, tolerability, pharmacokinetic(PK) profile, and anti-tumor efficacy of SKB445 for injection in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation, multicenter study to evaluate the safety, tolerability, PK characteristics, immunogenicity, and preliminary anti-tumor activity of SKB445 monotherapy in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the ICF: age between 18 -75 years, male or female.
2. subjects with histologically or cytologically confirmed locally advanced or metastatic solid tumors who have failed/are intolerant/ineligible to or do not have standard therapy, and have at least one measurable lesion meeting Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
3. Eastern Cooperative Oncology Group (ECOG) score of 0 to 1.
4. Expected survival ≥ 3 months.
5. Subjects with adequate organ and bone marrow function confirmed by laboratory results
6. Subjects of childbearing potential (male or female) must use effective medical contraception during the study
7. Ability to understand and willingness to sign ICF, and will be able to comply with the protocol-specified visits and relevant procedures.

Exclusion Criteria:

1. Has received anti-tumor therapy, including chemotherapy, targeted therapy, tumor immunotherapy, and traditional Chinese medicinal products with anti-tumor indications, within 4 weeks prior to the first dose or within 5 half-lives of known drugs (whichever is shorter).
2. Has had major surgery within 4 weeks prior to the first dose.
3. Has known history of allergy to any component of SKB445 or SKB445.
4. Has a known previous or concurrent other malignancies within 3 years prior to first dose.
5. Presence of active central nervous system (CNS) metastases.
6. Has uncontrolled or severe cardiovascular disease.
7. Has uncontrolled systemic diseases.
8. Has human immunodeficiency virus (HIV) infection; has any active viral hepatitis.
9. Subjects with a known history of psychiatric illness or drug abuse that would preclude the subject from complying with the study.
10. Has prior autologous/allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
11. Has any other conditions such as medical history, treatment and laboratory abnormalities that may confound the study results, interfere with the subject's compliance, or impair the subject's interests, as assessed by the investigator or the sponsor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects achieving Dose-limiting toxicity (DLT) | From date of initial dose until up to 21 days for treatment
  DLT is defined as an adverse event (AE) that meets protocol defined DLT criteria during cycle 1 and is at least possibly related to study drug.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 3 years
  The sum of the number of cases with Complete Response (CR) and Partial Response (PR) in all treated tumor patients (CR + PR) divided by the total number of cases.
Progression Free Survival (PFS) | Up to 3 years
  Time from start of treatment to progression of disease (PD) or death, whichever occurs first, in patients with tumors.
Duration of Response (DOR) | Up to 3 years
  Time from the start of the first assessment of CR or PR in tumor patients to PD or death due to any reason.
Overall Survival (OS) | Up to 3 years
  Time from start of treatment to death due to any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Shandong First Medical University, Jinan, Shandong, China